CLINICAL TRIAL: NCT04606563
Title: Host Response Mediators in Coronavirus (COVID-19) Infection - Is There a Protective Effect of Losartan and Other ARBs on Outcomes of Coronavirus Infection?
Acronym: ARBs CORONA II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMC recommendation due to futility
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jim Russell, Study Wide Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-01984
Record Dates: First submitted 2020-10-27; First posted 2020-10-28 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: ARBs; angiotensin II type 1 receptor blocker; ACEi; acute respiratory distress syndrome; COVID-19; coronavirus; multisite; Global; Canada; Acute kidney injury; acute cardiac injury; shock
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome; Coronavirus Infections; Acute Kidney Injury; Shock | interventions — Losartan; Valsartan; azilsartan; candesartan; candesartan cilexetil; eprosartan; Irbesartan; olmesartan; Olmesartan Medoxomil; Telmisartan

STUDY DESIGN:
Masking Description: Our RCT uses blinded randomization and a usual care control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan) (Experimental): Patients will initially receive initial dose of oral ARBs, increased to higher dose after 24 hours and then increased to a max dose after another 24 hours, dependent on tolerance. Patient will remain at dose for duration of hospital (max of 3 months if still hospitalized). Tolerance is defined as having no severe adverse events 24 hours after the first dose. Investigators and/or attending physicians discretion may dictate that dose will not be increased, at which point dose will stay at initial or higher dose.
  Interventions: Drug: Losartan; Drug: Valsartan; Drug: Azilsartan; Drug: Candesartan; Drug: Eprosartan; Drug: Irbesartan; Drug: Olmesartan; Drug: Telmisartan
- Usual Care Control (No Intervention): Usual care for duration of hospitalization for up to 3 months if still hospitalized. Due to the lack of clinical guidance from this emergent disease, this may vary dependent on Institution and/or country

INTERVENTIONS:
Drug: Losartan — Oral losartan 25 mg, stepped up to 50 mg and then up to 100 mg peak dose, as tolerated.
  Other Names: Cozaar
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Valsartan — Oral Valsartan 40 mg, stepped up to 80 mg and then up to 160 mg peak dose, as tolerated.
  Other Names: Diovan
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Azilsartan — Oral Azilsartan 40 mg, and stepped up to 80 mg.
  Other Names: Edarbi
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Candesartan — Oral Candesartan 8 mg, stepped up to 16 mg and then up to 32 mg peak dose, as tolerated.
  Other Names: Atacand
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Eprosartan — Oral Eprosartan 400 mg, stepped up to 600 mg and then up to 800 mg peak dose, as tolerated.
  Other Names: Teventen
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Irbesartan — Oral Irbesartan 75 mg, stepped up to 150 mg and then up to 300 mg peak dose, as tolerated.
  Other Names: Avapro
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Olmesartan — Oral Olmesartan 10 mg, stepped up to 20 mg and then up to 40 mg peak dose, as tolerated.
  Other Names: Olmetec
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)
Drug: Telmisartan — Oral Azilsartan 40 mg, and stepped up to 80 mg.
  Other Names: Micardis
  Arms: ARBs (Losartan, Valsartan, Azilsartan, Candesartan, Eprosartan, Irbesartan, Olmesartan, Telmisartan)

SUMMARY:
SARS-CoV-2 is a member of a class of viruses: angiotensin converting enzyme 2 (ACE2)-binding viruses that study calls "ABVs". The World Health Organization (WHO) and others are performing randomized controlled trials (RCTs) of vaccines and novel antivirals to address SARS-CoV-2 directly. However, the critical illness complications of COVID-19 are caused in part by SARS-CoV-2's binding and inhibiting ACE2 and the consequent host response.

ACE 2 is the receptor for H1N1, H5N1, and SARS-CoV-2. After binding ACE2, SARS-CoV-2 is endocytosed, and surface ACE2 is down-regulated, increasing angiotensin II (ATII a potent vasoconstrictor) in COVID-19. The original ARBs limits lung injury in murine influenza H7N9 and decreases viral titre and RNA.

Study has a unique opportunity to complement vaccine and anti-viral RCTs with an RCT modulating the host response using an angiotensin II type 1 receptor blocker (ARBs) to decrease the mortality of hospitalized COVID-19 patient.

DETAILED DESCRIPTION:
PURPOSE: There is clinical equipoise around the safety and efficacy of ARBs in COVID-19, but there are few RCTs of ARBs in COVID-19. Guo and colleagues' meta-analysis showed that ARBs/ACE inhibitor use was associated with decreased mortality. Our structured literature review (Cheng et al., submitted) shows that SARS-CoV-2 and other viruses that bind ACE2 cause acute cardiac injury in nearly 50% of cases. Safety concerns of ARBs in COVID-19 arise because ARBs increase cardiac ACE2, potentially increasing SARS-CoV-2 cellular uptake and worsening outcomes. On the other hand, ARBs block the effects of excess angiotensin II and could be beneficial. Our proposed ARBs CORONA II Phase 3 RCT will establish whether ARBs can decrease mortality in hospitalized COVID-19 patients.

HYPOTHESIS:

Primary - ARBs (losartan, valsartan, azilsartan, candesartan, eprosartan, irbesartan, olmesartan, telmisartan) decreases mortality and are safe in hospitalized COVID-19 infected adults compared to standard of care.

Secondary - ACE pathway proteins (ATI, AT1-7, ATII, ACE and ACE2 levels), cytokines and metabolomics/proteomics predict mortality and efficacy of ARBs in hospitalized COVID19 adults.

RESEARCH DESIGN: Study will assess ARBs (losartan, valsartan, azilsartan, candesartan, eprosartan, irbesartan, olmesartan, telmisartan) (see 6.3 Intervention for more) vs. usual care for safety and efficacy in decreasing organ dysfunction and mortality of hospitalized adults with COVID-19. Dr. Srinivas Murthy and Dr Rob Fowler, co-investigators herein and PIs of the CATCO RCT in Canada, Dr. John Marshall, co-investigator herein and PI of REMAPCAP, and Dr. Russell have coordinated alignment by allowing co-enrollment and harmonization of data and sample collection and primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized
* Must be first admission of COVID-19, not re-admission
* Primary reason for hospitalization or prolonged hospitalization is because of acute COVID-19 diagnosis
* Adults 18 years of age or greater
* Laboratory-proven COVID-19 within 14 days prior to hospital admission

Exclusion Criteria:

* Hypotension (SAP < 100 mmHg or DAP < 50 mmHg or MAP < 65 mmHg)
* Hyperkalemia (> 5.5 mmol/l)
* Acute kidney injury (urine output < 0.5 ml/kg/hr and new creatinine > 200 mmol/l, or increase > 100 mmol/l, or GFR < 30 ml/min)
* Use of aliskiren in patients with diabetes mellitus (type 1 or type 2) or moderate-severe renal impairment (GFR less than 60mL/min)
* Use of ARB/ACEi within 7 days of presentation
* Pregnant or breastfeeding
* Have a known allergy to ARBs or any component of the drug product
* Have written legal document to withhold life-sustaining (patients not wishing to receive Cardiopulmonary Resuscitation (CPR) can participate if other medical treatments will be given)
* Have signed a Do No Resuscitate (DNR) Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Survival status

SECONDARY OUTCOMES:
Hospital Mortality | up to 6 months
  Survival status
ICU Admission | up to 6 months
  Location within hospital (ICU or wards)
Days alive and free of vasopressors, ventilation, and renal replacement therapy | up to 14 days
  Survival and ICU support status
SOFA score | 28 days
  Sequential Organ Failure Assessment (SOFA) score
Acute cardiac injury | 6 months
  Use of inotropic agents and increase(s) of of troponin and/or NT-proBNP from admission level
Severe adverse events | 6 months
  Severe adverse effects of ARBs and mortality
Mortality | at 1, 3 and 6 months
  Survival status

CONTACTS AND LOCATIONS:
Overall Officials: James A Russell, MD, Principal Investigator — University of British Columbia; Karen Tran, MD, Principal Investigator — University of British Columbia
Locations (13):
- Canada (12):
  - University of Calgary - Foothills, Calgary, Alberta
  - Royal Jubilee Hospital, Nanaimo, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health, Saint Catharines, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - CHU de Québec - Université Laval, Laval, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- Centre Hospitalier Universitaire d'Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran KC, Asfar P, Cheng M, Demiselle J, Singer J, Lee T, Sweet D, Boyd J, Walley K, Haljan G, Sharif O, Geri G, Auchabie J, Quenot JP, Lee TC, Tsang J, Meziani F, Lamontagne F, Dubee V, Lasocki S, Ovakim D, Wood G, Turgeon A, Cohen Y, Lebas E, Goudelin M, Forrest D, Teale A, Mira JP, Fowler R, Daneman N, Adhikari NKJ, Gousseff M, Leroy P, Plantefeve G, Rispal P, Courtois R, Winston B, Reynolds S, Birks P, Bienvenu B, Tadie JM, Talarmin JP, Ansart S, Russell JA; ARBs CORONA II Team. Effects of Losartan on Patients Hospitalized for Acute COVID-19: A Randomized Controlled Trial. Clin Infect Dis. 2024 Sep 26;79(3):615-625. doi: 10.1093/cid/ciae306. PMID 39325643